CLINICAL TRIAL: NCT05223478
Title: Randomized, Parallel Arm, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) to Reverse Pharmacologically Induced Mydriasis in Healthy Pediatric Subjects
Brief Title: Nyxol (0.75% Phentolamine Ophthalmic Solution) to Reverse Pharmacologically-Induced Mydriasis in Pediatric Subjects
Acronym: MIRA-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPI-NYXRMP-303 (MIRA-4)
Record Dates: First submitted 2021-12-16; First posted 2022-02-04 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Mydriasis; Dilation
Keywords: Nyxol; Pharmacologically Induced Mydriasis; Dilation; Pediatrics; Phentolamine; Mydriasis; Phenylephrine; Tropicamide; Paremyd
MeSH Terms: conditions — Mydriasis; Dilatation, Pathologic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentolamine Ophthalmic Solution 0.75% (Active Comparator): One drop of study medication in each eye.
  Interventions: Drug: Phentolamine Ophthalmic Solution 0.75%
- Phentolamine Ophthalmic Solution Vehicle (Placebo Comparator): One drop of study medication in each eye.
  Interventions: Drug: Phentolamine Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: Phentolamine Ophthalmic Solution 0.75% — 0.75% phentolamine ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol®; Nyxol
  Arms: Phentolamine Ophthalmic Solution 0.75%
Drug: Phentolamine Ophthalmic Solution Vehicle — Phentolamine Ophthalmic Solution Vehicle
  Arms: Phentolamine Ophthalmic Solution Vehicle

SUMMARY:
The objectives of this study are:

* To evaluate the safety of Nyxol in pediatric subjects
* To evaluate the efficacy of Nyxol to expedite the reversal of pharmacologically induced mydriasis in pediatric subjects The Sponsor intends to use this study to evaluate Nyxol in pediatric subjects aged 3 to 11 for the indication "the treatment of pharmacologically induced mydriasis produced by adrenergic (phenylephrine) or parasympatholytic (tropicamide) agents, or a combination thereof."

DETAILED DESCRIPTION:
This is a randomized, parallel-arm, double-masked, placebo-controlled study in approximately 20 randomized pediatric subjects evaluating the safety and efficacy of Nyxol in pediatric subjects with pharmacologically induced mydriasis with three dilating agents (e.g., phenylephrine, tropicamide, and Paremyd). Pediatric subjects will be recruited for the study into 2 age groups as follows:1) 3 to 5 years of age: 10 subjects 2) 6 to 11 years of age: 10 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or premenstrual females 3 to 11 years of age
2. Ability to comply with all protocol-mandated procedures independently and to attend all scheduled office visits
3. Parent/Legal guardian willing to give written informed consent to participate in this study. Children aged 7 to 11 years to provide signed assent form, as well as a separate parental/legal guardian consent.

Exclusion Criteria:

1. Clinically significant ocular disease as deemed by the Investigator(eg, amblyopia, congenital cataract, congenital glaucoma) that might interfere with the study
2. Unwilling or unable to discontinue use of contact lenses at screening until study completion
3. Unwilling or unable to suspend use of topical medication at screening until study completion
4. Ocular trauma or ocular surgery within the 6 months prior to screening
5. Use of any topical prescription or over-the-counter (OTC)ophthalmic medications of any kind within 7 days of screening
6. Recent or current evidence of ocular infection or inflammation in either eye (such as current evidence of clinically significant blepharitis, conjunctivitis, or keratitis). Subjects must be symptom-free for at least 7 days prior to screening
7. Closed or very narrow-angle that in the Investigator's opinion is potentially occludable if the subject's pupil is dilated
8. History of any traumatic (surgical or nonsurgical) or non-traumatic condition affecting the pupil or iris
9. Known allergy, hypersensitivity, or contraindication to any component of the phentolamine ophthalmic solution or to any component of the mydriatic agents or vehicle formulation

   Systemic:
10. Known hypersensitivity or contraindication to α- and/or β-adrenoceptor antagonists
11. Clinically significant systemic disease (eg, uncontrolled diabetes, cancer, hepatic, renal, endocrine, or cardiovascular disorders) that in the opinion of the Investigator could interfere with the study
12. Subjects with learning disabilities that in the opinion of the investigator could interfere with the study
13. Initiation of treatment with or any changes to the current dosage, drug, or regimen of any systemic adrenergic or cholinergic drugs within 7 days prior to screening or during the study(Appendix 4)
14. Participation in any investigational study within 30 days prior to screening

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Slonim, MD, Study Director — Oculos Development Services
Locations (2):
- United States (2):
  - Clinical Site 1, Longwood, Florida
  - Clinical Site 2, Athens, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 12 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (2.74) | 5.8 (2.66) | 6.3 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Safety Measurements
Description: Study Eye Change from Baseline (-1 Hour) Conjunctival Hyperemia Grading; Cornea and Contact Lens Research Unit (CCLRU scale) Grades range from 0 to 3, with 3 being considered the most severe.
Time Frame: 0 Minutes, 90 Minutes, 3 Hours, 24 Hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
score on a scale
  0 Minutes | 0.3 (0.65) | -0.2 (0.58)
  90 Minutes | 1.6 (0.50) | 0.0 (0.43)
  3 Hours | 1.1 (0.54) | -0.1 (0.29)
  24 Hours | 0.1 (0.30) | -0.2 (0.58)

2. Primary Outcome: Vital Signs
Description: Change from Screening Heart Rate
Time Frame: 3 Hours, 24 Hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
beats per minute
  3 Hours | -1.1 (7.92) | -2.0 (14.24)
  24 Hours | -2.5 (10.10) | -3.5 (12.69)

3. Primary Outcome: Vital Signs
Description: Change from Screening Blood Pressure (Systolic)
Time Frame: 3 Hours, 24 Hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
mmHg
  3 Hours | -4.6 (8.91) | -0.8 (12.39)
  24 Hours | -2.8 (7.48) | -5.8 (6.98)

4. Primary Outcome: Safety Measurement
Description: Study Eye Change from Baseline (-1 Hour) in Best Corrected Distance Visual Acuity
Time Frame: 0 Minutes, 3 Hours, 24 Hours
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
letters
  0 Minutes | -1.2 (1.66) | -0.3 (1.23)
  3 Hours | 1.2 (1.89) | 0.1 (0.67)
  24 Hours | 1.5 (1.97) | 0.7 (1.15)

5. Primary Outcome: Change From Screening Blood Pressure (Diastolic)
Time Frame: 3 Hours, 24 Hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
mmHg
  3 Hours | -2.4 (9.72) | 1.0 (15.68)
  24 Hours | -1.1 (11.63) | -3.8 (7.96)

6. Secondary Outcome: Efficacy Measurement: Pupil Diameter
Description: Percentage of Subjects Returning to ≤ 0.2 mm from Baseline (-1 hour) Pupil Diameter (Study Eye)
Time Frame: 90 Minutes, 3 Hours, and 24 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
Participants
  90 Minutes | 7 | 3
  3 Hours | 9 | 4
  24 Hours | 10 | 6

7. Secondary Outcome: Efficacy Measurement: Pupil Diameter
Description: Change (in mm) in Pupil Diameter from Max Pupil Dilation (0 minutes) (Study Eye)
Time Frame: 90 Minutes, 3 Hours, and 24 Hours
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
millimeters
  90 Minutes | -1.475 (0.7188) | -0.378 (0.4473)
  3 Hours | -2.031 (0.6919) | -0.723 (0.6470)
  24 Hours | -2.005 (1.2841) | -1.44 (1.2891)

8. Secondary Outcome: Efficacy Measurement: Pupil Diameter
Description: Time (Hours) to Return to ≤ 0.2 mm from Baseline (-1 Hour) Pupil Diameter (Time-savings Analysis) (Study Eye)
Time Frame: Up to 24 Hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 11 | 12
hours | 2.95 (2.564) | 5.54 (3.078)

ADVERSE EVENTS:
Time Frame: 2 Days
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT05223478/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT05223478/SAP_001.pdf